CLINICAL TRIAL: NCT00050817
Title: A Phase III, Multicenter, Multinational, Randomized, Parallel Group, Double-blind Trial of Clopidogrel Versus Placebo in High-risk Patients Aged 45 Years and Older, at Risk of Atherothrombotic Events, and Who Are Receiving Background Therapy Including Low-dose ASA.
Brief Title: Clopidogrel for High Atherothrombotic Risk and Ischemic Stabilization, Management and Avoidance (CHARISMA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4505
Record Dates: First submitted 2002-12-20; First posted 2002-12-23 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Arteriosclerosis
Keywords: Embolism
MeSH Terms: conditions — Arteriosclerosis; Embolism | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: clopidogrel (SR25990)

SUMMARY:
RATIONALE:

* Atherothrombosis is a progressive and generalized vascular disease resulting in events leading to myocardial infarction (heart attack), stroke, and vascular death.
* In patients at risk for this disease, it is characterized by an unpredictable, sudden disruption of atherosclerotic plaques, which may lead to total occlusion of artery due to formation of a clot. The use of aspirin (blood thinner agent) for reducing those major ischemic events is either indicated, or recommended by international guidelines. However, aspirin fails to prevent a high percentage of such life-threatening events. Therefore, more effective blood thinning therapy may provide additional clinical benefit to such patients.
* The results of the CURE trial in patients with unstable angina demonstrate the additional benefit of long-term treatment (up to one year) with clopidogrel, (a blood thinner agent), when administered in combination with standard therapy including aspirin. The purpose of CHARISMA is to investigate whether a similar clinical benefit of clopidogrel may apply to a broad population of high-risk patients receiving low-dose aspirin therapy. Such population includes patients with previous cardiovascular, neurovascular or peripheral arterial manifestations of atherothrombosis and patients with combinations of recognized risk factors for atherosclerosis.

OBJECTIVES:

* To assess the efficacy of clopidogrel 75 mg once-daily by comparison with a placebo, in preventing cardiovascular morbidity/mortality. The study will compare the efficacy of the two regimens in preventing the occurrence of major cardiovascular complications (stroke, heart attack, cardiovascular death) in high-risk patients who are otherwise receiving low-dose aspirin therapy (75-162 mg daily).
* To evaluate the safety of clopidogrel in this population, and more specifically the incidence of fatal or severe bleeding (as per GUSTO definition), in order to estimate the global benefit of clopidogrel in this patient population.

DETAILED DESCRIPTION:
TREATMENTS:

* Clopidogrel (Plavix® and/or Iscover®) is an agent inhibiting platelet aggregation involved in clot formation. Each tablet contains 75mg of clopidogrel. A matching placebo of clopidogrel is an inactive substance that looks similar to the active clopidogrel tablet.

TREATMENT PLAN:

* There will be two treatment groups; one will receive clopidogrel 75 mg (1 tablet qd), the second matching placebo of clopidogrel (1 tablet qd). These study drugs will be administered on top of low-dose aspirin (75-162 mg qd) systematically prescribed to such patients. In addition, patients enrolled in CHARISMA will be managed as appropriate for their risk factors for atherosclerosis: eg. high blood pressure, high cholesterol, diabetes…etc.

PRIMARY ENDPOINT:

* Combined endpoint of cardiovascular mortality, stroke, acute myocardial infarction.

STUDY EXECUTION:

* Some 7,600 patients per group will be recruited within two years. Patients will be observed over a maximum of 3.5 years.

STUDY TERRITORY:

* Approximately 900 sites throughout North/South America, Europe, Asia, Australia, and South Africa.

ELIGIBILITY:
INCLUSION:

Be at least 45 years old and comply with at least one of the four categories of inclusion criteria:

* Combination of atherothrombotic risk factors (2 major or 3 minor or 1 major + 2 minor risk factors among those listed below)

Major atherothrombotic risk factors

* Type I or II diabetes (under drug therapy)
* Diabetic nephropathy
* Ankle brachial index (ABI) < 0.9
* Asymptomatic carotid stenosis >= 70%
* At least one carotid plaque as evidenced by intima-media thickness (IMT)

Minor atherothrombotic risk factors

* Systolic blood pressure (SBP) >= 150 mmHg, despite appropriate therapy for at least 3 months
* Primary hypercholesterolemia
* Current smoking > 15 cigarettes per day
* Male >= 65 years
* Female >= 70 years

and/or

* Documented cerebrovascular disease (TIA or IS within 5 years) and/or
* Documented coronary artery disease (stable angina with documented multivessel coronary disease, previous documented MI, multivessel PCI or CABG within 1 year, multivessel CABG older than 1 year associated with current angina) and/or
* Documented symptomatic PAD

EXCLUSION:

* Absolute indication for the use of clopidogrel, high-dose aspirin (>162 mg), NSAIDs, or oral anti-thrombotic drugs
* Absolute contraindication to the use of clopidogrel or aspirin
* Clinical conditions likely to interfere with follow-up leading to inability to complete the trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15603 (Actual)
Dates: Start 2002-10; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of myocardial infarction,stroke or cardiovascular death.

SECONDARY OUTCOMES:
severe bleeding

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (32):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States
- Sanofi-aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-aventis Administrative Office, Macquarie Park, Australia
- Sanofi-aventis Administrative Office, Vienna, Austria
- Sanofi-aventis Administrative Office, Diegem, Belgium
- Sanofi-aventis Administrative Office, São Paulo, Brazil
- Sanofi-aventis Administrative Office, Laval, Canada
- Sanofi-aventis Administrative Office, Santiago, Chile
- Sanofi-aventis Administrative Office, Prague, Czechia
- Sanofi-aventis Administrative Office, Hørsholm, Denmark
- Sanofi-aventis Administrative Office, Helsinki, Finland
- Sanofi-aventis Administrative Office, Paris, France
- Sanofi-aventis Administrative Office, Berlin, Germany
- Sanofi-aventis Administrative Office, Athens, Greece
- Sanofi-aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-aventis Administrative Office, Budapest, Hungary
- Sanofi-aventis Administrative Office, Milan, Italy
- Sanofi-aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-aventis Administrative Office, México, Mexico
- Sanofi-aventis Administrative Office, Gouda, Netherlands
- Sanofi-aventis Administrative Office, Lysaker, Norway
- Sanofi-aventis Administrative Office, Warsaw, Poland
- Sanofi-aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-aventis Administrative Office, Moscow, Russia
- Sanofi-aventis Administrative Office, Singapore, Singapore
- Sanofi-aventis Administrative Office, Midrand, South Africa
- Sanofi-aventis Administrative Office, Barcelona, Spain
- Sanofi-aventis Administrative Office, Bromma, Sweden
- Sanofi-aventis Administrative Office, Geneva, Switzerland
- Sanofi-aventis Administrative Office, Taipei, Taiwan
- Sanofi-aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] Bhatt DL, Fox KA, Hacke W, Berger PB, Black HR, Boden WE, Cacoub P, Cohen EA, Creager MA, Easton JD, Flather MD, Haffner SM, Hamm CW, Hankey GJ, Johnston SC, Mak KH, Mas JL, Montalescot G, Pearson TA, Steg PG, Steinhubl SR, Weber MA, Brennan DM, Fabry-Ribaudo L, Booth J, Topol EJ; CHARISMA Investigators. Clopidogrel and aspirin versus aspirin alone for the prevention of atherothrombotic events. N Engl J Med. 2006 Apr 20;354(16):1706-17. doi: 10.1056/NEJMoa060989. Epub 2006 Mar 12. PMID 16531616
- [Result] Bhatt DL, Pare G, Eikelboom JW, Simonsen KL, Emison ES, Fox KA, Steg PG, Montalescot G, Bhakta N, Hacke W, Flather MD, Mak KH, Cacoub P, Creager MA, Berger PB, Steinhubl SR, Murugesan G, Mehta SR, Kottke-Marchant K, Lincoff AM, Topol EJ; CHARISMA Investigators. The relationship between CYP2C19 polymorphisms and ischaemic and bleeding outcomes in stable outpatients: the CHARISMA genetics study. Eur Heart J. 2012 Sep;33(17):2143-50. doi: 10.1093/eurheartj/ehs059. Epub 2012 Mar 26. PMID 22450429
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Bangalore S, Bhatt DL, Steg PG, Weber MA, Boden WE, Hamm CW, Montalescot G, Hsu A, Fox KA, Lincoff AM. beta-blockers and cardiovascular events in patients with and without myocardial infarction: post hoc analysis from the CHARISMA trial. Circ Cardiovasc Qual Outcomes. 2014 Nov;7(6):872-81. doi: 10.1161/CIRCOUTCOMES.114.001073. Epub 2014 Sep 30. PMID 25271049
- [Derived] Berger PB, Bhatt DL, Fuster V, Steg PG, Fox KA, Shao M, Brennan DM, Hacke W, Montalescot G, Steinhubl SR, Topol EJ; CHARISMA Investigators. Bleeding complications with dual antiplatelet therapy among patients with stable vascular disease or risk factors for vascular disease: results from the Clopidogrel for High Atherothrombotic Risk and Ischemic Stabilization, Management, and Avoidance (CHARISMA) trial. Circulation. 2010 Jun 15;121(23):2575-83. doi: 10.1161/CIRCULATIONAHA.109.895342. Epub 2010 Jun 1. PMID 20516378
- [Derived] Steinhubl SR, Bhatt DL, Brennan DM, Montalescot G, Hankey GJ, Eikelboom JW, Berger PB, Topol EJ; CHARISMA Investigators. Aspirin to prevent cardiovascular disease: the association of aspirin dose and clopidogrel with thrombosis and bleeding. Ann Intern Med. 2009 Mar 17;150(6):379-86. doi: 10.7326/0003-4819-150-6-200903170-00006. PMID 19293071
- [Derived] Mak KH, Bhatt DL, Shao M, Haffner SM, Hamm CW, Hankey GJ, Johnston SC, Montalescot G, Steg PG, Steinhubl SR, Fox KA, Topol EJ. The influence of body mass index on mortality and bleeding among patients with or at high-risk of atherothrombotic disease. Eur Heart J. 2009 Apr;30(7):857-65. doi: 10.1093/eurheartj/ehp037. Epub 2009 Feb 20. PMID 19233855
- [Derived] Eikelboom JW, Hankey GJ, Thom J, Bhatt DL, Steg PG, Montalescot G, Johnston SC, Steinhubl SR, Mak KH, Easton JD, Hamm C, Hu T, Fox KA, Topol EJ; Clopidogrel for High Atherothrombotic Risk and Ischemic Stabilization, Management and Avoidance (CHARISMA) Investigators. Incomplete inhibition of thromboxane biosynthesis by acetylsalicylic acid: determinants and effect on cardiovascular risk. Circulation. 2008 Oct 21;118(17):1705-12. doi: 10.1161/CIRCULATIONAHA.108.768283. Epub 2008 Oct 6. PMID 18838564
- [Derived] Bhatt DL, Flather MD, Hacke W, Berger PB, Black HR, Boden WE, Cacoub P, Cohen EA, Creager MA, Easton JD, Hamm CW, Hankey GJ, Johnston SC, Mak KH, Mas JL, Montalescot G, Pearson TA, Steg PG, Steinhubl SR, Weber MA, Fabry-Ribaudo L, Hu T, Topol EJ, Fox KA; CHARISMA Investigators. Patients with prior myocardial infarction, stroke, or symptomatic peripheral arterial disease in the CHARISMA trial. J Am Coll Cardiol. 2007 May 15;49(19):1982-8. doi: 10.1016/j.jacc.2007.03.025. Epub 2007 Apr 11. PMID 17498584